CLINICAL TRIAL: NCT04222400
Title: Feasibility and Comparison of the Impact of Different Frailty Assessment Tools on the Outcome of Ventricular Assist Device Implantation and Heart Transplantation
Brief Title: Comparison of Different Frailty Assessment Tools
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Heart Institute (Other)
Collaborators: The German Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FrailtyVAD-Tx
Record Dates: First submitted 2019-08-08; First posted 2020-01-10 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
Keywords: Advanced Heart Failure; Ventricular Assist Device; Heart Transplantation; Frailty; Sarcopenia; Bioelectrical Impedance Analysis; Muscle Mass
MeSH Terms: conditions — Heart Failure; Frailty; Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transplantation (Active Comparator): Frailty assessment before, after and 6 month after surgery
  Interventions: Diagnostic Test: Frailty Assessment
- VAD Implantation (Active Comparator): Frailty assessment before, after and 6 month after surgery
  Interventions: Diagnostic Test: Frailty Assessment

INTERVENTIONS:
Diagnostic Test: Frailty Assessment — Bioelectrical Impedance Analysis 6 Minute Walk Test Grip Strength Questionnaires Muscle Mass Evaluation via CT

SUMMARY:
Feasibility and Comparison of the Impact of different Frailty Assessment Tools on the Outcome of Ventricular Assist Device Implantation and Heart Transplantation in advanced heart failure patients

DETAILED DESCRIPTION:
Comparison of the feasibility and results of the following frailty assessment tools in advanced heart failure patients treated with ventricular assist device Implantation or awaiting heart transplantation in Eurotransplant-Status "high urgency":

* Evaluation of the muscle mass in the preoperative CT-Scan
* Bioelectrical Impedance Analysis
* 6 Minute Walk Test
* Grip Strength Measurement
* Questionnaires: EQ5D-5L, Rockwood Frailty Scale

The assessment will be conducted prior to surgery, after surgery and at 6 Month Follow-up

ELIGIBILITY:
Inclusion Criteria:

* Planned VAD Implantation/ HU-Status awaiting Heart Transplantation
* Signature on Informed Consent

Exclusion Criteria:

* < 18 years old
* Informed consent not possible/not signed
* Pregnancy/Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of not performed tests due to clinical concerns/inability of the patient (feasibility and safety) | Pre-operative measurements,
  Number of patients, who were not able to perform tests and reasons
Incidence of not performed tests due to clinical concerns/inability of the patient (feasibility and safety) | post-operative measurements in the week before discharge (average 4 weeks)
  Number of patients, who were not able to perform tests and reasons
Incidence of not performed tests due to clinical concerns/inability of the patient (feasibility and safety) | 6 Month Follow-up
  Number of patients, who were not able to perform tests and reasons
Impact of frailty estimated by the different frailty assessment tools on the outcome 6 month mortality and/or prolonged ventilation time | After 6 Month
  Combined Endpoint: Endpoint is met if the Patient dies within 6 month after surgery and/or needed of a prolonged ventilation time of >95h during the ICU stay after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Felix Schoenrath, MD, Principal Investigator — German Heart Center Berlin
Locations (1):
- German Heart Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roehrich L, Sundermann SH, Just IA, Kopp Fernandes L, Stein J, Solowjowa N, Mulzer J, Mueller M, Hummel M, Knierim J, Potapov E, Falk V, Schoenrath F. Comparison of feasibility and results of frailty assessment methods prior to left ventricular assist device implantation. ESC Heart Fail. 2022 Apr;9(2):1038-1049. doi: 10.1002/ehf2.13764. Epub 2022 Jan 6. PMID 34994094